CLINICAL TRIAL: NCT00939003
Title: A Multicenter Study of the Efficacy and Safety of the Human Anti-TNF Monoclonal Antibody Adalimumab in Subjects With Axial Spondyloarthritis
Brief Title: Study of Adalimumab in Patients With Axial Spondyloarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M10-791; 2009-010643-14 (EudraCT Number)
Record Dates: First submitted 2009-07-10; First posted 2009-07-14 (Estimated); Results first posted 2012-03-06 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Axial Spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Adalimumab (Experimental)
  Interventions: Biological: Adalimumab
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo
- Open-label Adalimumab (Experimental)
  Interventions: Biological: Open-label Adalimumab

INTERVENTIONS:
Biological: Adalimumab — 40 mg every other week up to Week 12
  Other Names: ABT-D2E7; Humira
  Arms: Adalimumab
Biological: Placebo — Placebo every other week up to Week 12
  Arms: Placebo
Biological: Open-label Adalimumab — 40 mg every other week, Week 12 through Week 156
  Other Names: ABT-D2E7; Humira
  Arms: Open-label Adalimumab

SUMMARY:
This study will evaluate how well adalimumab works in the short and long term in patients with axial spondyloarthritis who are not diagnosed as having either ankylosing spondylitis or psoriatic arthritis.

DETAILED DESCRIPTION:
This is a Phase 3, placebo-controlled, double-blind randomized study with an open-label phase designed to evaluate the efficacy and safety of adalimumab 40 mg administered every other week in adult patients with active axial spondyloarthritis (SpA) who are not diagnosed with ankylosing spondylitis, psoriasis, or psoriatic arthritis and who have had an inadequate response or intolerance to one or more nonsteroidal anti-inflammatory drugs (NSAIDs) or had a contraindication to NSAIDs. Participants receive adalimumab or placebo for 12 weeks during the double-blind phase of the study. Following the double-blind phase, all remaining participants enter the open-label phase of the study in which they receive open-label adalimumab for up to 144 weeks. Efficacy endpoints include the Assessment of Spondyloarthritis International Society (ASAS) response criteria for patients with SpA. These response criteria were used to determine participants who were responders. ASAS response involves evaluations in the following 4 domains: participant's global assessment of disease activity, pain, function, and inflammation. The patient's global assessment of disease activity score is assessed using a 100 millimeter (mm) visual analog scale (VAS; 0 for no disease activity to 100 for severe disease activity). Pain is represented as a total back pain score and is assessed using a 100 mm VAS (0 for no pain to 100 for most severe pain). Function score is represented as the Bath Ankylosing Spondylitis (AS) Functional Index (BASFI) 100 mm VAS score (average of the ability to perform 10 activities, each scored as 0 for easy to 100 for impossible). Inflammation is determined using the morning stiffness overall level score (0 for none to 10 for very severe) and duration score (0 for 0 hours to 10 for ≥ 2 hours) of the Bath AS Disease Activity Index (BASDAI) (mean of these items #5 and #6 scores). In addition, the BASDAI is used as an efficacy endpoint. The BASDAI is used by the participant to assess his/her disease activity. Using VAS scales, the participant answers 6 questions pertaining to symptoms experienced over the past week. For 5 questions (levels of: fatigue/tiredness; AS neck, back, or hip pain; pain/swelling; discomfort at areas tender to touch or pressure; and morning stiffness), the response scale is 0 (none) to 10 (very severe). For 1 question (duration of morning stiffness), the response scale is 0 (0 hours) to 10 (≥ 2 or more hours).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with inadequate response to >/= 1 non-steroidal anti-inflammatory drugs (NSAIDs)
* Chronic back pain with onset < 45 years of age
* Magnetic resonance imaging (MRI) indicating active sacroiliitis or positive human leukocyte antigen-B27 (HLA-B27) blood test in addition to meeting spondyloarthritis clinical criteria
* Negative purified protein derivative (PPD) test and chest x-ray performed at Baseline visit must be negative
* Ability to administer subcutaneous injections
* General good health otherwise

Exclusion Criteria:

* Prior anti-tumor necrosis factor (TNF) therapy
* Psoriasis or psoriatic arthritis
* Fulfillment of modified New York criteria for ankylosing spondylitis
* Recent infection requiring treatment
* Significant medical events or conditions that may put patients at risk for participation
* Females who are pregnant or breast-feeding or considering becoming pregnant during the study
* History of cancer, except successfully treated skin cancer
* Recent history of drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2009-07; Primary Completion 2011-02 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aileen L Pangan, MD, Study Director — AbbVie
Locations (38):
- United States (9):
  - Site Reference ID/Investigator# 21250, Birmingham, Alabama
  - Site Reference ID/Investigator# 21249, Colorado Springs, Colorado
  - Site Reference ID/Investigator# 21245, Denver, Colorado
  - Site Reference ID/Investigator# 21246, Wheaton, Maryland
  - Site Reference ID/Investigator# 26582, Duncansville, Pennsylvania
  - Site Reference ID/Investigator# 21241, Wyomissing, Pennsylvania
  - Site Reference ID/Investigator# 21243, Dallas, Texas
  - Site Reference ID/Investigator# 21248, Houston, Texas
  - Site Reference ID/Investigator# 21247, Seattle, Washington
- Australia (3):
  - Site Reference ID/Investigator# 22342, Brisbane
  - Site Reference ID/Investigator# 21223, Kogarah
  - Site Reference ID/Investigator# 21222, Maroochydore
- Belgium (4):
  - Site Reference ID/Investigator# 21225, Genk
  - Site Reference ID/Investigator# 21224, Ghent
  - Site Reference ID/Investigator# 26544, Gilly
  - Site Reference ID/Investigator# 27382, Merksem
- Canada (4):
  - Site Reference ID/Investigator# 21229, Edmonton
  - Site Reference ID/Investigator# 21226, Sainte-Foy, Quebec
  - Site Reference ID/Investigator# 21227, St. John's
  - Site Reference ID/Investigator# 21228, Toronto
- Czechia (4):
  - Site Reference ID/Investigator# 21231, Brno
  - Site Reference ID/Investigator# 26882, Pardubice
  - Site Reference ID/Investigator# 21230, Prague
  - Site Reference ID/Investigator# 26883, Uherské Hradiště
- France (4):
  - Site Reference ID/Investigator# 21263, Boulogne-Billancourt
  - Site Reference ID/Investigator# 21262, Chambray-les-Tour
  - Site Reference ID/Investigator# 21261, Orléans
  - Site Reference ID/Investigator# 22343, Paris
- Germany (4):
  - Site Reference ID/Investigator# 21266, Berlin
  - Site Reference ID/Investigator# 21267, Erlangen
  - Site Reference ID/Investigator# 21264, Herne
  - Site Reference ID/Investigator# 21265, Munich
- Netherlands (2):
  - Site Reference ID/Investigator# 21285, Amsterdam
  - Site Reference ID/Investigator# 21284, Leiden
- Spain (3):
  - Site Reference ID/Investigator# 21282, A Coruña
  - Site Reference ID/Investigator# 21283, Barcelona
  - Site Reference ID/Investigator# 21281, Córdoba
- Site Reference ID/Investigator# 21289, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Derived] van der Heijde D, Sieper J, Maksymowych WP, Lambert RG, Chen S, Hojnik M, Anderson JK, Pangan AL. Clinical and MRI remission in patients with nonradiographic axial spondyloarthritis who received long-term open-label adalimumab treatment: 3-year results of the ABILITY-1 trial. Arthritis Res Ther. 2018 Mar 27;20(1):61. doi: 10.1186/s13075-018-1556-5. PMID 29587851
- [Derived] van der Heijde D, Sieper J, Maksymowych WP, Brown MA, Lambert RG, Rathmann SS, Pangan AL. Spinal inflammation in the absence of sacroiliac joint inflammation on magnetic resonance imaging in patients with active nonradiographic axial spondyloarthritis. Arthritis Rheumatol. 2014 Mar;66(3):667-73. doi: 10.1002/art.38283. PMID 24574227
- [Derived] Sieper J, van der Heijde D, Dougados M, Mease PJ, Maksymowych WP, Brown MA, Arora V, Pangan AL. Efficacy and safety of adalimumab in patients with non-radiographic axial spondyloarthritis: results of a randomised placebo-controlled trial (ABILITY-1). Ann Rheum Dis. 2013 Jun;72(6):815-22. doi: 10.1136/annrheumdis-2012-201766. Epub 2012 Jul 7. PMID 22772328
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 192 participants were enrolled at 37 study sites in Australia, Belgium, Canada, the Czech Republic, France, Germany, the Netherlands, Spain, the United Kingdom, and the US. Due to Investigator non-compliance with protocol requirements, 1 study site was closed; the 7 participants enrolled at this site were excluded from efficacy analyses.
Groups:
- Placebo: Participants received placebo every other week for 12 weeks during the double-blind period and then received adalimumab 40 mg subcutaneously every other week for up to 144 weeks during the open-label period.
- Adalimumab: Participants received adalimumab 40 mg subcutaneously every other week for 12 weeks during the double-blind period and then received adalimumab 40 mg subcutaneously every other week for up to 144 weeks during the open-label period.
Period: Double-blind Treatment Period
Arm/Group | Placebo | Adalimumab
Started | 97 | 95
Completed | 95 | 91
Not Completed | 2 | 4
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Pregnancy | 0 | 1
Not completed — MRI Not Diagnostic | 1 | 1
Period: Open-label Treatment Period
Arm/Group | Placebo | Adalimumab
Started | 95 | 91
Completed | 66 | 62
Not Completed | 29 | 29
Not completed — Adverse Event | 4 | 8
Not completed — Withdrawal by Subject | 14 | 7
Not completed — Lack of Efficacy | 6 | 9
Not completed — Pregnancy | 1 | 1
Not completed — Exclusion Criteria | 1 | 0
Not completed — Site Closure | 3 | 4

BASELINE CHARACTERISTICS:
Population: Full analysis set, defined as all participants who received at least one dose of blinded study drug excluding seven participants from one site due to investigator non-compliance.
Groups:
- Double-blind Adalimumab: Participants received adalimumab 40 mg subcutaneously every other week for 12 weeks during the double-blind period and then received adalimumab 40 mg subcutaneously every other week for up to 144 weeks during the open-label period.
- Total: Total of all reporting groups
Arm/Group | Placebo | Double-blind Adalimumab | Total
Number analyzed (Participants) | 94 | 91 | 185
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (10.39) | 37.6 (11.29) | 38.0 (10.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 47 | 101
  Male | 40 | 44 | 84

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving an Assessment of Spondyloarthritis International Society (ASAS) 40 Response
Description: ASAS40 response was defined as improvement of ≥ 40% relative to Baseline and absolute improvement of ≥ 20 units (on a scale from 0 to 100) in ≥ 3 of the following 4 domains with no deterioration (defined as a net worsening of > 0 units on a scale from 0 to 100) in the potential remaining domain:
  * Patient's Global Assessment of disease activity, measured on a visual analog scale (VAS) from 0 (none) to 100 (severe);
  * Pain, measured by the total back pain VAS from 0 (no pain) to 100 (most severe);
  * Function, measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) which consists of 10 items assessing participants' ability to perform activities on a VAS ranging from 0 (easy) to 100 (impossible);
  * Inflammation, measured by the mean of the 2 morning stiffness-related Bath AS Disease Activity Index (BASDAI) VAS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Time Frame: Baseline and Week 12
Population: Full analysis set. Participants with missing data at Week 12 were counted as non-responders (non-responder imputation).
Measure: Number; unit: participants
Groups:
- Double-blind Placebo: Double-blind placebo every other week for 12 weeks
- Double-blind Adalimumab: Double-blind adalimumab 40 mg subcutaneously every other week for 12 weeks
Arm/Group | Double-blind Placebo | Double-blind Adalimumab
Number analyzed (Participants) | 94 | 91
participants | 14 | 33
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Adalimumab; Test type: Superiority or Other; p < 0.001, Chi-squared

2. Secondary Outcome: Number of Participants Achieving an Assessment of Spondyloarthritis International Society (ASAS) 20 Response
Description: ASAS20 response was defined as improvement of ≥ 20% relative to Baseline and absolute improvement of ≥ 10 units (on a scale from 0 to 100) in ≥ 3 of the following 4 domains with no deterioration (defined as a change for the worse of ≥ 20% and net worsening of ≥ 10 units) in the potential remaining domain:
  * Patient's Global Assessment of disease activity, measured on a visual analog scale (VAS) from 0 (none) to 100 (severe);
  * Pain, measured by the total back pain VAS from 0 (no pain) to 100 (most severe);
  * Function, measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) which consists of 10 items assessing participants' ability to perform activities on a VAS ranging from 0 (easy) to 100 (impossible);
  * Inflammation, measured by the mean of the 2 morning stiffness-related Bath AS Disease Activity Index (BASDAI) VAS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Time Frame: Baseline and Week 12
Population: Full analysis set; Non-responder imputation performed.
Measure: Number; unit: participants
Arm/Group | Double-blind Placebo | Double-blind Adalimumab
Number analyzed (Participants) | 94 | 91
participants | 29 | 47
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Adalimumab; Test type: Superiority or Other; p = 0.004, Chi-squared

3. Secondary Outcome: Number of Participants Achieving a Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) 50 Response
Description: The Bath Ankylosing Spondylitis (AS) Disease Activity Index assesses disease activity by asking the participant to answer 6 questions (each on a 10 cm VAS) pertaining to symptoms experienced for the past week. For 5 questions (level of fatigue/tiredness, level of AS neck, back or hip pain, level of pain/swelling in joints, other than neck, back or hips, level of discomfort from any areas tender to touch or pressure, and level of morning stiffness), the response is from 0 (none) to 10 (very severe); for Question 6 (duration of morning stiffness), the response is from 0 (0 hours) to 10 (≥ 2 hours). The overall BASDAI score ranges from 0 to 10 cm. Lower scores indicate less disease activity. BASDAI50 is a 50% improvement from Baseline in BASDAI score.
Time Frame: Baseline and Week 12
Population: Full analysis set; Non-responder imputation performed.
Measure: Number; unit: participants
Arm/Group | Double-blind Placebo | Double-blind Adalimumab
Number analyzed (Participants) | 94 | 91
participants | 14 | 32
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Adalimumab; Test type: Superiority or Other; p = 0.001, Chi-squared

4. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Physical Component Summary Score
Description: The Medical Outcome Study Short Form 36-Item Health Survey, Version 2 (SF-36) is a self-administered instrument that measures the impact of disease on overall quality of life. The SF-36 consists of 36 questions in 8 domains (limitations in physical functioning due to health problems; limitations in usual role because of physical health problems; bodily pain; general health perceptions; vitality; limitations in social functioning because of physical or emotional problems; limitations in usual role due to emotional problems; and general mental health). Two component scores can be summarized: physical and mental; domains 1-4 comprise the physical component summary of the SF-36. A transformed summary score is calculated ranging from 0 to 100 where higher scores indicate a higher level of functioning. A positive change from Baseline score indicates an improvement.
Time Frame: Baseline and Week 12
Population: Full analysis set with available data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind Placebo | Double-blind Adalimumab
Number analyzed (Participants) | 93 | 91
units on a scale | 2.0 (7.04) | 5.5 (8.98)
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Adalimumab; Test type: Superiority or Other; p = 0.001, ANCOVA; ANCOVA model adjusting for Baseline value with treatment as a factor

5. Secondary Outcome: Number of Participants Achieving ASAS Partial Remission
Description: ASAS partial remission is an absolute score of < 20 units on a 0 to 100 scale for each of the four following domains:
  * Patient's Global Assessment of disease activity, measured on a visual analog scale (VAS) from 0 (none) to 100 (severe);
  * Pain, measured by the total back pain VAS from 0 (no pain) to 100 (most severe);
  * Function, measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) which consists of 10 items assessing participants' ability to perform activities on a VAS ranging from 0 (easy) to 100 (impossible);
  * Inflammation, measured by the mean of the 2 morning stiffness-related Bath AS Disease Activity Index (BASDAI) VAS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Time Frame: Week 12
Population: Full analysis set; Non-responder imputation performed.
Measure: Number; unit: participants
Arm/Group | Double-blind Placebo | Double-blind Adalimumab
Number analyzed (Participants) | 94 | 91
participants | 5 | 15
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Adalimumab; Test type: Superiority or Other; p = 0.014, Chi-squared

6. Other Pre Specified Outcome: Number of Participants Reporting Adverse Events
Description: Adverse events were collected at designated study visits for all participants who received at least 1 dose of study drug. The number of participants experiencing any adverse event (serious and non-serious) is summarized.
Time Frame: Through Week 12
Population: All participants who received at least 1 dose of study drug. For the double-blind phase of the study, adverse events are reported through Week 12.
Measure: Number; unit: participants
Arm/Group | Double-blind Placebo | Double-blind Adalimumab
Number analyzed (Participants) | 97 | 95
participants | 57 | 55

7. Other Pre Specified Outcome: Number of Participants With Blood Hematology or Chemistry Values Common Toxicity Criteria Grade ≥ 3
Description: Blood was collected for analysis at designated study visits; hematology and chemistry results were provided by a central laboratory. The number of participants with an abnormal laboratory result (higher then upper normal limit or lower than lower normal limit) meeting Common Toxicity Criteria (CTC) of Grade 3 or higher is summarized.
Time Frame: Through Week 12
Population: All participants who received at least 1 dose of study drug. Results for the double-blind phase phase of the study are reported through Week 12.
Measure: Number; unit: participants
Arm/Group | Double-blind Placebo | Double-blind Adalimumab
Number analyzed (Participants) | 97 | 95
participants | 6 | 4

8. Secondary Outcome: Number of Participants Achieving an ASAS5/6 Response
Description: ASAS5/6 response is a 20% improvement in five out of the following six domains:
  * Patient's Global Assessment of disease activity, measured on a visual analog scale (VAS) from 0 (none) to 100 (severe);
  * Pain, measured by the total back pain VAS from 0 (no pain) to 100 (most severe);
  * Function, measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) which consists of 10 items assessing participants' ability to perform activities on a VAS ranging from 0 (easy) to 100 (impossible);
  * Inflammation, measured by the mean of the 2 morning stiffness-related Bath AS Disease Activity Index (BASDAI) VAS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none) to 10 (very severe/2 hours or more duration).
  * Spinal mobility, measured from the lateral lumbar flexion score of the Bath AS Metrology Index (BASMI) on a scale from 0 (best mobility) to 10 (worst mobility);
  * C-reactive protein level (lower levels indicate less inflammation).
Time Frame: Baseline and Week 12
Population: Full analysis set; Non-responder imputation performed.
Measure: Number; unit: participants
Arm/Group | Double-blind Placebo | Double-blind Adalimumab
Number analyzed (Participants) | 94 | 91
participants | 6 | 28
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Adalimumab; Test type: Superiority or Other; p < 0.001, Chi-squared

9. Secondary Outcome: Change From Baseline in Disability Index of Health Assessment Questionnaire Modified for the Spondyloarthropathies (HAQ-S)
Description: Health Assessment Questionnaire modified for spondyloarthropathies (HAQ-S) is a self-reported measure to assess the physical function and health-related quality of life. The Disability Index (DI) of HAQ-S is calculated as the mean of the following 8 category scores (range: 0 [without any difficulty] to 3 [unable to do]): Dressing and Grooming, Rising, Eating, Walking, Hygiene, Reach, Grip, and Activities. Five additional items in the functional status measure were included in the HAQ-S, including carrying heavy packages, sitting for long periods, able to work at a flat topped table, and (if the participant had a driver's license or a car) able to look in the rear view mirror and able to turn head to drive in reverse. The overall score ranges from 0 (no disability) to 3 (three very severe, high-dependency disability). Negative mean changes from Baseline in the overall score indicate improvement.
Time Frame: Baseline and Week 12
Population: Full analysis set; participants with non-missing Baseline and at least one non-missing post-baseline values were included. Last observation carried forward was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind Placebo | Double-blind Adalimumab
Number analyzed (Participants) | 94 | 91
units on a scale | -0.1 (0.42) | -0.3 (0.49)
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Adalimumab; Test type: Superiority or Other; p = 0.027, ANCOVA; ANCOVA model adjusting for Baseline value with treatment as a factor

10. Secondary Outcome: Change From Baseline in High-Sensitivity C-Reactive Protein (hsCRP)
Description: C-reactive protein (CRP) is considered an efficacy variable for the axial spondyloarthritis indication. It is a general marker of inflammation that is sensitive to acute changes in inflammatory response. Higher levels indicate more inflammation.
Time Frame: Baseline and Week 12
Population: Full analysis set; participants with non-missing Baseline and at least one non-missing post-baseline value were included. Last observation carried forward was used.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Double-blind Placebo | Double-blind Adalimumab
Number analyzed (Participants) | 73 | 70
mg/L | -0.3 (6.39) | -4.7 (12.32)
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Adalimumab; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA model adjusting for Baseline value with treatment as a factor

11. Secondary Outcome: Change From Baseline in Spondyloarthritis Research Consortium of Canada (SPARCC) Magnetic Resonance Imaging (MRI) Score for Sacroiliac Joints
Description: Six consecutive sacroiliac (SI) joint image coronal slices representing the largest proportion of the synovial compartment of the SI joints were assessed for edema, intensity and depth of edema using SPARCC scoring.
  Each SI joint (left and right) was divided into quadrants for a total of 8 SI scoring locations. Each quadrant was scored for the presence (1) or absence (0) of edema; the maximum score is 8 per slice and maximum score for 6 SI joint slices is 48.
  Intensity of edema: A score of 1 was assigned for each SI joint (left and right) if an intense signal was seen in any quadrant of that joint for each slice. The maximum score is 2 per slice and 12 for 6 slices.
  A lesion was graded as deep (score of 1) if there was homogeneous and unequivocal increase in signal extending over a depth of at least 1 cm from the articular surface of the SI joint in any quadrant. The maximum score per slice is 2 and for 6 slices 12.
  The total maximum score for all SI joints across 6 slices is 72.
Time Frame: Baseline and Week 12
Population: Full analysis set; participants with non-missing Baseline and non-missing post-baseline value were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind Placebo | Double-blind Adalimumab
Number analyzed (Participants) | 84 | 84
units on a scale | -0.6 (6.19) | -3.2 (8.34)
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Adalimumab; Test type: Superiority or Other; p = 0.003, ANCOVA; ANCOVA model adjusting for Baseline value with treatment as a factor

12. Secondary Outcome: Change From Baseline in SPARCC MRI Score for the Spine
Description: Six discovertebral units (DVU) representing the 6 most abnormal DVUs, and 3 consecutive sagittal slices at each DVU representing the most abnormal slices for that DVU were selected for scoring. Each DVU was divided into 4 quadrants and scored for the presence (1) or absence (0) of edema. The maximum score is 12 per DVU. The maximum score is 72 for 6 DVUs.
  If edema was present in at least 1 quadrant of a DVU slice, it was scored for intensity and depth of the edema representing that slice:
  A score of 1 was assigned if an intense signal was seen in any quadrant on a DVU slice. The maximum score for intensity per slice is 1, per DVU is 3 and for 6 DVUs is 18.
  A lesion was graded as deep (score of 1) if there was homogeneous and unequivocal increase in signal extending over a depth of at least 1 cm from the surface of the endplate in any quadrant. The maximum score per slice is 1, for a DVU is 3 and for 6 DVUs is 18.
  The total maximum SPARCC score for all 6 DVUs is 108.
Time Frame: Baseline and Week 12
Population: Full analysis set; participants with non-missing Baseline and non-missing post-baseline value were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-blind Placebo | Double-blind Adalimumab
Number analyzed (Participants) | 82 | 85
units on a scale | -0.2 (3.35) | -1.8 (4.51)
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Adalimumab; Test type: Superiority or Other; p = 0.001, ANCOVA; ANCOVA model adjusting for Baseline value with treatment as a factor

13. Other Pre Specified Outcome: Number of Participants Achieving an ASAS20 Response During the Open-label Period
Description: as for outcome 2
Time Frame: Baseline and Weeks 52, 104, and 156
Population: Full analysis set participants with available data at each time point (as indicated by N)
Measure: Number; unit: participants
Arm/Group | Placebo | Adalimumab
Number analyzed (Participants) | 94 | 91
participants
  Week 52 (N=78, 72) | 59 | 57
  Week 104 (N=74, 64) | 59 | 53
  Week 156 (N=64, 58) | 53 | 48

14. Other Pre Specified Outcome: Number of Participants Achieving an ASAS40 Response During the Open-label Period
Description: ASAS40 response was defined as improvement of ≥ 40% relative to Baseline and absolute improvement of ≥ 20 units (on a scale from 0 to 100) in ≥ 3 of the following 4 domains with no deterioration (defined as a net worsening of > 0 units on a scale of 0 to 100) in the potential remaining domain:
  * Patient's Global Assessment of disease activity, measured on a visual analog scale (VAS) from 0 (none) to 100 (severe);
  * Pain, measured by the total back pain VAS from 0 (no pain) to 100 (most severe);
  * Function, measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) which consists of 10 items assessing participants' ability to perform activities on a VAS ranging from 0 (easy) to 100 (impossible);
  * Inflammation, measured by the mean of the 2 morning stiffness-related Bath AS Disease Activity Index (BASDAI) VAS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Time Frame: Baseline and Weeks 52, 104, and 156
Population: Full analysis set participants with available data at each time point (indicated by N)
Measure: Number; unit: participants
Arm/Group | Placebo | Adalimumab
Number analyzed (Participants) | 94 | 91
participants
  Week 52 (N=78, 72) | 50 | 42
  Week 104 (N=74, 64) | 51 | 38
  Week 156 (N=64, 58) | 44 | 37

15. Other Pre Specified Outcome: Number of Participants Achieving a BASDAI50 Response During the Open-label Period
Description: as for outcome 3
Time Frame: Baseline and Weeks 52, 104, and 156
Population: Full analysis set participants with available data at each time point (indicated by N)
Measure: Number; unit: participants
Arm/Group | Placebo | Adalimumab
Number analyzed (Participants) | 94 | 91
participants
  Week 52 (N=78, 72) | 52 | 42
  Week 104 (N=74, 64) | 50 | 40
  Week 156 (N=64, 58) | 46 | 39

ADVERSE EVENTS:
Time Frame: Twelve weeks during the double blind period and up to Week 156 during the open-label period.
Groups:
- Double-blind Placebo: Participants received placebo every other week for 12 weeks during the double-blind period.
- Double-blind Adalimumab: Participants received adalimumab 40 mg subcutaneously every other week for 12 weeks during the double-blind period.
- Any Adalimumab: Participants who received any dose of adalimumab during the 12-week double-blind period or during the 144-week open-label period.
Arm/Group | Double-blind Placebo | Double-blind Adalimumab | Any Adalimumab
Serious Adverse Events (participants affected / at risk) | 1/97 | 3/95 | 33/190
Other Adverse Events (participants affected / at risk) | 32/97 | 42/95 | 152/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Placebo (N=97) | Double-blind Adalimumab (N=95) | Any Adalimumab (N=190)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 0 | 0 | 1
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 1
GOITRE (Endocrine disorders) | 0 | 0 | 1
MACULAR DEGENERATION (Eye disorders) | 0 | 0 | 1
OSCILLOPSIA (Eye disorders) | 0 | 0 | 1
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 0
STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 1
VOMITING (Gastrointestinal disorders) | 1 | 0 | 0
CHEST PAIN (General disorders) | 0 | 0 | 1
CHILLS (General disorders) | 1 | 0 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 1
PYREXIA (General disorders) | 1 | 0 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 0 | 1
HEPATITIS ACUTE (Hepatobiliary disorders) | 0 | 1 | 1
BURSITIS INFECTIVE (Infections and infestations) | 0 | 0 | 1
CELLULITIS (Infections and infestations) | 0 | 0 | 2
DISSEMINATED TUBERCULOSIS (Infections and infestations) | 0 | 0 | 1
DIVERTICULITIS (Infections and infestations) | 0 | 0 | 1
PILONIDAL CYST (Infections and infestations) | 0 | 0 | 1
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 | 0 | 1
SINUSITIS (Infections and infestations) | 0 | 0 | 1
TONSILLITIS (Infections and infestations) | 0 | 0 | 1
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 1
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 | 0 | 1
LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
LUPUS-LIKE SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
PERIARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
TENDON CALCIFICATION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 0 | 0 | 2
MIGRAINE (Nervous system disorders) | 0 | 0 | 1
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
COMPLETED SUICIDE (Psychiatric disorders) | 0 | 0 | 1
SUICIDE ATTEMPT (Psychiatric disorders) | 0 | 0 | 1
BREAST DYSPLASIA (Reproductive system and breast disorders) | 0 | 1 | 1
MENORRHAGIA (Reproductive system and breast disorders) | 0 | 0 | 1
VAGINAL PROLAPSE (Reproductive system and breast disorders) | 0 | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
ABORTION INDUCED (Surgical and medical procedures) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Placebo (N=97) | Double-blind Adalimumab (N=95) | Any Adalimumab (N=190)
CONJUNCTIVITIS (Eye disorders) | 0 | 0 | 6
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 2 | 9
CONSTIPATION (Gastrointestinal disorders) | 3 | 1 | 2
DIARRHOEA (Gastrointestinal disorders) | 7 | 4 | 18
NAUSEA (Gastrointestinal disorders) | 7 | 7 | 13
ASTHENIA (General disorders) | 2 | 3 | 7
FATIGUE (General disorders) | 0 | 3 | 14
INJECTION SITE ERYTHEMA (General disorders) | 0 | 3 | 6
INJECTION SITE PAIN (General disorders) | 3 | 1 | 2
INJECTION SITE REACTION (General disorders) | 0 | 4 | 11
PYREXIA (General disorders) | 0 | 2 | 8
BRONCHITIS (Infections and infestations) | 2 | 1 | 31
CYSTITIS (Infections and infestations) | 0 | 0 | 7
GASTROENTERITIS (Infections and infestations) | 3 | 2 | 11
INFLUENZA (Infections and infestations) | 0 | 2 | 9
NASOPHARYNGITIS (Infections and infestations) | 3 | 11 | 52
ORAL HERPES (Infections and infestations) | 0 | 2 | 6
PHARYNGITIS (Infections and infestations) | 0 | 3 | 15
RHINITIS (Infections and infestations) | 2 | 2 | 9
SINUSITIS (Infections and infestations) | 2 | 1 | 18
TONSILLITIS (Infections and infestations) | 2 | 1 | 9
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 3 | 19
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 7
VAGINAL INFECTION (Infections and infestations) | 1 | 0 | 6
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 0 | 0 | 7
CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 7
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 6
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 1 | 6
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 6
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 1 | 11
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 13
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 9
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 6
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 1 | 7
SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 2 | 2 | 37
SPONDYLOARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 8
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 6
HEADACHE (Nervous system disorders) | 3 | 6 | 19
ANXIETY (Psychiatric disorders) | 0 | 0 | 11
DEPRESSION (Psychiatric disorders) | 0 | 2 | 7
INSOMNIA (Psychiatric disorders) | 0 | 2 | 9
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 8
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 9
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 1 | 6
RASH (Skin and subcutaneous tissue disorders) | 2 | 2 | 6
HYPERTENSION (Vascular disorders) | 2 | 0 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.